CLINICAL TRIAL: NCT06176794
Title: A Crossover Study of Patients With Heart Failure to Compare Natriuretic Effects of Immediate Release Torsemide vs. Extended Release Torsemide Over 12 Hours After Dosing
Brief Title: Immediate Release Torsemide Versus Extended Release Torsemide After Salty Meal
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Issues with recruitment
Sponsor: Sarfez Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SAR065-224; GM0016563 (Other Grant/Funding Number: Sarfez Pharmaceuticals)
Record Dates: First submitted 2023-12-11; First posted 2023-12-20 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Tablets

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Extended release torsemide (Experimental)
  Interventions: Drug: Immediate release torsemide 20mg tablet; Drug: Extended release torsemide 24mg tablet
- Immediate release torsemide (Active Comparator)
  Interventions: Drug: Immediate release torsemide 20mg tablet; Drug: Extended release torsemide 24mg tablet

INTERVENTIONS:
Drug: Immediate release torsemide 20mg tablet — Subjects will receive approximately one week of daily immediate release 20mg torsemide (plus daily placebo of 24mg extended release torsemide) and one week of daily extended release 24mg torsemide (plus daily placebo of 20mg immediate release torsemide) with no gap in between. Subjects will be randomly assigned to immediate-release torsemide-first arm versus extended-release torsemide-first arm and at the end of the initial one-week period, they will be switched to the other intervention. Subjects will consume only the provided meals with standardized amount of sodium content throughout the study period.
Drug: Extended release torsemide 24mg tablet — Subjects will receive approximately one week of daily immediate release 20mg torsemide (plus daily placebo of 24mg extended release torsemide) and one week of daily extended release 24mg torsemide (plus daily placebo of 20mg immediate release torsemide) with no gap in between. Subjects will be randomly assigned to immediate-release torsemide-first arm versus extended-release torsemide-first arm and at the end of the initial one-week period, they will be switched to the other intervention. Subjects will consume only the provided meals with standardized amount of sodium content throughout the study period.

SUMMARY:
The goal of this randomized double-blind crossover study is to assess whether a morning dose of the extended release torsemide has a better efficacy than the ordinary immediate release torsemide to induce renal sodium excretion after a salty lunch in patients with stable heart failure. The main questions it aims to answer are:

* Are the amounts of excreted sodium in the urine during the 2- and 6-hours' time period after a morning dose of extended release torsemide different from the amounts after the immediate release torsemide.
* Are the amounts of excreted sodium in the urine during the 2- and 6-hours' time period after a salty lunch, which will be consumed approximately 6 hours following a morning dose of extended release torsemide, different from the amounts after the immediate release torsemide.
* Is the amount of excreted sodium in the urine during the 24 hours' time period after a salty lunch, which will be consumed approximately 6 hours following a morning dose of extended release torsemide, different from the amount after the immediate release torsemide.

Participants will be asked to:

* Start taking daily immediate release or extended release torsemide tablets that is provided to them.
* Eat the meals with standard contents of sodium that is provided to them and avoid other meals, drinks (except for water) and snacks for the duration of the study.
* Collect urine for 24 hours, after approximately one week of the initiation of the study medication.
* Go to the clinical research center the day that the 24-hour urine collection is finished and stay there throughout the day to receive standard meals and to have blood and urine samples collected.
* Switch torsemide pills to the new one that will be dispensed to them at the clinical research center. If they were taking the immediate release torsemide during the first part, then they will be given the sustained release torsemide and vice versa. The study is double blind; therefore, the subjects, study coordinators, and investigators are unaware of whether each subject is on immediate release torsemide first or on extended release torsemide first.
* Collect urine for an additional 12 hours after leaving the clinical research center to be sent to the clinical research center the next morning.
* Continue to take the provided meals and to avoid other meals, drinks (except for water) and snacks.
* Again, collect urine for 24 hours, after approximately one week, take that to the clinical research center when the 24-hour collection is completed and stay there throughout the day to receive standard meals and to have blood and urine samples collected.
* Collect urine for an additional 12 hours to be sent to the clinical research center the next morning.

Researchers will compare the amount of sodium excretion when each subject is taking immediate release torsemide versus the time that the same subject is taking extended release torsemide.

DETAILED DESCRIPTION:
Sarfez Inc has developed an extended release formulation of torsemide, whose effect lasts for several hours after the dosing. The purpose of this study is to assess whether a morning dose of the extended release torsemide has a better efficacy than the ordinary immediate release torsemide to induce renal sodium excretion after a salty lunch.

This is a randomized double-blind crossover study of the patients with stable heart failure, who are on a stable dose of a loop diuretic. During the study period, the participants' loop diuretics will be replaced by the equivalent dose of immediate release/extended release torsemide and they will receive standardized meals throughout the study period. After a "week" of taking a morning dose of each of the two torsemide formulations, serial urinary sodium measurements following a salty lunch will be compared between the time that the subject was taking the immediate release vs. the time period that the subject was taking the extended release torsemide as a single morning dose.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman over the age of 18 years.
* Willing and able to sign the informed consent.
* A clinical diagnosis of chronic HF that is considered by patient's cardiologist/physician to be stable over the one-month period prior to randomization.
* Receiving a stable dose of furosemide of 40mg or 80mg total per day (or equivalent doses of torsemide or bumetanide) for at least 30 days prior to randomization.
* Optimum volume status determined by experienced physician.
* Able to consume a diet containing approximately 3 grams of Na+ daily.
* No anticipated changes in HF medications during the study period.

Exclusion Criteria:

* Requirement for a diuretic other than furosemide, bumetanide or torsemide except for spironolactone, eplerenone, finerenone, or SGLT2 inhibitors, given in stable dose for > 2 weeks before randomization and during the study.
* Known non-adherence to medication intake or salt restriction.
* Myocardial infarction, stroke, transient ischemic attack, acute kidney injury or acute HF requiring admission to hospital within the last 30 days prior to randomization.
* Severe / symptomatic lung disease or respiratory symptoms distinct from HF.
* Urinary incontinence or inability to empty bladder with a post-void residual volume >100 ml.
* Uncontrolled diabetes mellitus or uncontrolled hypertension.
* Estimated GFR < 30 ml/min/1.72m2 of body surface area.
* Use of any non-loop diuretic in the last 30 days prior to randomization, with the exception of a low dose MRA (e.g., spironolactone of 25-50 mg per day) or an SGLT2 inhibitor.
* History of flash pulmonary edema or amyloid cardiomyopathy.
* Requirement for a non-steroidal anti-inflammatory drug other than low dose aspirin (<200 mg daily)
* Refusal or inability to sign the informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2024-11-15 (Actual); Primary Completion 2025-03-25 (Actual); Study Completion 2025-03-25 (Actual)

PRIMARY OUTCOMES:
Cumulative Na+ excretion over 6 hours | 6 hours after lunch
  The primary outcome is the cumulative Na+ excretion over 6 hours after lunch.

SECONDARY OUTCOMES:
Fluid and Na+ excretion over the 6 hours | 6 hours after breakfast, 6 hours after lunch, and 24 hours
  Fluid and Na+ excretion over the 6 hours after breakfast, 6 hours after lunch, and 24 hours after dosing.
creatinine clearance | While in the study (approximately 2 weeks)
  Safety outcome
K+ excretion | While in the study (approximately 2 weeks)
  Safety outcome

CONTACTS AND LOCATIONS:
Overall Officials: Parta Hatamizadeh, MD, MPH, Principal Investigator — University of Florida
Locations (1):
- Division of Nephrology, Hypertension & Renal Transplantation, University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No